CLINICAL TRIAL: NCT06513767
Title: A Prospective, Multicentre, Single-group, Target-value Clinical Investigation Evaluating the Safety and Efficacy of Zirconia Ceramic Blocks for All-ceramic Dentures for Use in Dental Prostheses.
Brief Title: A Clinical Investigation to Evaluate the Safety and Efficacy of Zirconia Ceramic Blocks for Use in Dental Prostheses.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Kerui Medical Technology Co., Ltd (Other)
Collaborators: SHENZHEN XIANGTONG CO., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F2024-006-1
Record Dates: First submitted 2024-06-27; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Dental Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational group (Experimental): Use of the investigational device (zirconia dental ceramic) to perform dental restorations
  Interventions: Device: Zirconia Dental Ceramics

INTERVENTIONS:
Device: Zirconia Dental Ceramics — This investigation was conducted by enrolling subjects who met the enrolment criteria, using the investigational device (Zirconia Dental Ceramics) to perform dental prosthesess.

SUMMARY:
The goal of this clinical trial is to use the investigational device (Zirconia Dental Ceramics) to perform dental prosthesis in Patients with permanent teeth. The main question it aims to answer is:

Is the safety and efficacy of the investigational device (Zirconia Dental Ceramics) adequate to meet the requirements for clinical use?

Participants will use the investigational device (Zirconia Dental Ceramics) to perform dental prosthesis and then complete a 12-month follow-up after prostheses. During the follow-up period，participants will assess their satisfaction，while the investigator will assess the efficacy indices of prosthesis survival rate, prosthesis success rate and prosthesis quality.

DETAILED DESCRIPTION:
The study aims to provide clinical evidence for the use of the investigational product (zirconia dental ceramic) in dental restorations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. Patients with permanent teeth who were judged by the investigator to be expected to have dental prostheses using zirconia materials;
3. Subjects volunteered and signed an informed consent form.

Exclusion Criteria:

1. Allergy to zirconia ceramic materials or a history of extensive allergies;
2. Patients with oral mucosal ulcers;
3. Patients presents with a significant, uncontrolled, systemic disease, encompassing, but not limited to, cardiovascular disease, endocrine or metabolic disease, and immune system disease, among others;
4. Pregnant or breastfeeding, or those planning to become pregnant during the investigation period;
5. Participation in another clinical investigation within 3 months;
6. Patients with mental disorders and a lack of autonomy;
7. Meets other conditions that, in the opinion of the investigator, make participation in this clinical investigation inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Survival rate | Day 360
  Evaluation was performed by the treatment investigator based on the actual condition of the prostheses at the time of the subject's follow-up visit (in the event that multiple prostheses are present, the most unfavourable outcome is considered), and the appropriate medical images were retained. prostheses survival was calculated after completion of the D360 visit for all subjects.
  In the absence of interference from external factors (e.g., severe trauma), the prostheses are considered to be survivors if they remain in situ, with or without modification, throughout the observation period.

SECONDARY OUTCOMES:
Survival rate | Day 180
  Same as the Primary Outcome Measure
Success rate | Day 180, Day 360
  Evaluation was performed by the treatment investigator based on the actual condition of the prostheses at the time of the subject's follow-up visit (in the event that multiple prostheses are present, the most unfavourable outcome is considered.), and the corresponding medical images were retained. The relevant prostheses success rate was calculated after completion of the corresponding visits for all subjects.
  In the absence of interference from external factors (e.g., severe trauma), the prosthesis is considered a success if it is free of any complications over the entire observation period.
Prostheses quality | Day 0, Day 180, Day 360
  The quality of the prostheses was evaluated by the treatment investigator based on the actual condition of the prostheses at the time of the subject's follow-up visit and according to United States Public Health Services (USPHS) criteria.Each USPHS criterion was ranked on a scale of A to C, where A = excellent, B = good, C = unacceptable.
Subject satisfaction | Day 0, Day 180, Day 360
  The appearance and comfort of the prostheses were evaluated by the subjects according to their own subjective feelings. Visual Analogue Scales (VAS) was used to complete the satisfaction rating by themselves. That is, on a 10cm long scale, "0" represents the most satisfactory and "10" represents the most unbearable.